CLINICAL TRIAL: NCT06112847
Title: A Phase 2 Study of Epcoritamab and Lenalidomide (E-Len) in Patients With Previously Untreated Follicular Lymphoma (FL)
Brief Title: Lenalidomide and Epcoritamab for the Treatment of Previously Untreated Follicular Lymphoma
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Goal met
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22509; NCI-2023-08814 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22509 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Specimen Handling; Biopsy; Lenalidomide; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (lenalidomide and epcoritamab) (Experimental): Patients receive lenalidomide PO QD on days 1-21 of each cycle and epcoritamab SC on days 1, 8, 15, and 21 of cycles 1-3 and on day 1 of each subsequent cycle. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients may be re-treated with study treatment at any point during the follow-up period as long as they did not progress during treatment or stop due to unacceptable toxicity. Patients also undergo CT, PET/CT, or MRI as well as bone marrow biopsy throughout the trial. Patients undergo blood sample collection on trial and during follow-up.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Other: Electronic Health Record Review; Biological: Epcoritamab; Drug: Lenalidomide; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Other: Electronic Health Record Review — Ancillary studies
Biological: Epcoritamab — Given SC
  Other Names: Anti-CD20/CD3 Bispecific Antibody GEN3013; DuoBody-CD3xCD20; Epcoritamab-bysp; Epkinly; GEN 3013; GEN-3013; GEN3013
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This phase II trial tests how well lenalidomide and epcoritamab works in treating patients with follicular lymphoma that has not been previously treated. Although follicular lymphoma is incurable, prognosis has improved for both early and advanced stage disease, largely attributed to therapeutic advances. Lenalidomide may stimulate or suppress the immune system in different ways and stop cancer cells from growing and by preventing the growth of new blood vessels that cancer cells need to grow. Epcoritamab is a bispecific monoclonal antibody that binds to two different antigens (the part of the target that the antibody attaches to), at the same time. This dual action allows bispecific antibodies to improve target specificity by binding two antigens on the same cell to recruit and activate immune cells to kill cancer cells. Lenalidomide and epcoritamab, when given together, may be more effective in treating patients with follicular lymphoma than if they were given alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess efficacy (complete response [CR] rate) of epcoritamab and lenalidomide (E-Len) in patients with de novo follicular lymphoma (FL).

SECONDARY OBJECTIVES:

I. To further assess efficacy of the combination (objective response rate [ORR], progression free survival [PFS], duration of response).

II. To characterize the adverse event profile of the combination.

EXPLORATORY OBJECTIVES:

I. To characterize the T-cell population balance in patients treated with E-Len.

II. To evaluate the predictive role of genetic mutations on durability of response to E-Len (including m7 Follicular Lymphoma International Prognostic Index [FLIPI] score).

III. To evaluate minimal residual disease (MRD) dynamics on treatment.

OUTLINE:

Patients receive lenalidomide orally (PO) once daily (QD) on days 1-21 of each cycle and epcoritamab subcutaneously (SC) on days 1, 8, 15, and 21 of cycles 1-3 and on day 1 of each subsequent cycle. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients may be re-treated with study treatment at any point during the follow-up period as long as they did not progress during treatment or stop due to unacceptable toxicity. Patients also undergo computed tomography (CT), positron emission tomography (PET)/CT, or magnetic resonance imaging (MRI) as well as bone marrow biopsy throughout the trial. Patients undergo blood sample collection on trial and during follow-up.

After completion of study treatment, patients are followed for safety on days 7, 30, and 60, for active response every 6 months for up to 2 years, and then for survival every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Age: ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) ≤ 2
* Histologically confirmed previously untreated FL grade 1-3a, requiring therapy per Groupe d'Etude des Lymphomes Folliculaires (GELF) criteria
* Radiologically measurable lymphadenopathy (> 1.5 cm) or extranodal involvement (including spleen, bone marrow or other extranodal site)
* Without bone marrow involvement: Absolute neutrophil count (ANC) ≥ 1,000/mm^3 With bone marrow involvement: ANC ≥ 500/mm^3

  * NOTE: Growth factor is not permitted within 14 days of ANC assessment unless cytopenia is secondary to disease involvement
* Without bone marrow involvement: Platelets ≥ 50,000/mm^3 With bone marrow involvement: Platelets ≥ 25,000/mm^3

  * NOTE: Platelet transfusions are not permitted within 14 days of platelet assessment unless cytopenia is secondary to disease involvement.
* Total bilirubin ≤ 2 x upper limit of normal (ULN) (unless has Gilbert's disease)
* Aspartate aminotransferase (AST) ≤ 2.5 x ULN
* Alanine aminotransferase (ALT) ≤ 2.5 x ULN
* Creatinine clearance of ≥ 45 mL/min per 24 hour urine test or the Cockcroft-Gault formula or creatinine level < 1.5 mg/dL
* If not receiving anticoagulants: International normalized ratio (INR) OR prothrombin (PT) ≤ 1.5 x ULN
* If not receiving anticoagulants: Activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN
* Women of childbearing potential (WOCBP): Negative urine or serum pregnancy test

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential* to use an effective method of birth control (i.e., failure rate of < 1% per year) or abstain from heterosexual activity for the course of the study treatment period through at least 30 days after the last dose of lenalidomide, and 2 months after the last dose of epcoritamab, or 4 months after the last dose of tocilizumab (if applicable) whichever is longer

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from .menses for > 1 year (women only)

    * All study participants must be registered into the mandatory Revlimid Risk Evaluation and Mitigation Strategy (REMS)® program and be willing and able to comply with the requirements of the REMS program (including use of aspirin [ASA]/Food and Drug Administration [FDA] approved blood thinner)
    * Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS program

Exclusion Criteria:

* Prior therapeutic intervention with any anti-cancer agents; localized radiotherapy ≤ 20 Gy total dose is permissible if occurred ≥ 4 weeks prior to first dose of study medication.

  * Participants must have at least one non-irradiated target lesion
* Concurrent enrollment in another therapeutic investigational study
* Vaccinated with live vaccines within 4 weeks of the first dose of study drug
* Current evidence of central nervous system involvement by the lymphoma
* Grade 3b or transformed FL
* History of prior malignancy except:

  * Malignancy treated with curative intent and no known active disease present for ≥ 2 years prior to initiation of therapy on current study
  * Adequately treated non-melanoma skin cancer or lentigo maligna (melanoma in situ) without evidence of disease
  * Asymptomatic prostate cancer managed with "watch and wait" strategy or hormonal therapy
* Uncontrolled active systemic infection
* Absolute lymphocyte count > 5,000/uL
* Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection. Patients with past HBV infection (defined as negative hepatitis B virus surface protein antigen [HbsAg] and positive hepatitis B core antibody [HbcAb]) are eligible if HBV deoxyribonucleic acid (DNA) is undetectable. Patients who are positive for HCV antibody are eligible if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA). Testing to be done only in patients suspected of having infections or exposures
* Known active human immunodeficiency virus (HIV) infection. Subjects who have an undetectable or unquantifiable HIV viral load with CD4 > 200 and are on highly active antiretroviral therapy (HAART) medication are allowed. Testing to be done only in patients suspected of having infections or exposures
* Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months of screening
* Females only: Pregnant or breastfeeding or intending to become pregnant during the study or within 6 months after the final dose of all study drugs

  * Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to initiation of study drug
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2024-01-24 (Actual); Primary Completion 2026-07-17 (Estimated); Study Completion 2026-07-17 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) rate | Up to 2 years
  Defined as the proportion of response evaluable patients who achieve a complete response according to Lugano criteria on study before any documented disease progression or any subsequent non-Hodgkin lymphoma (NHL) treatment. Disease assessment will be performed by positron emission tomography (PET)-computed tomography (CT), CT, magnetic resonance imaging and/or bone marrow biopsy. PET-CT and CT results will be read by a radiologist and investigator response assessment will be performed. CR rate will be estimated along with the 95% exact binomial confidence interval.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 2 years
  Toxicity will be evaluated by Common Terminology Criteria for Adverse Events version 5 AE terms and grades. Observed toxicities will be summarized by type, severity, and attribution.
Overall response rate (ORR) | Up to 2 years
  The proportion of response evaluable patients who achieve CR or partial response (PR) according to Lugano 2016 guidelines on study before any documented disease progression or any subsequent NHL treatment. ORR will be estimated along with the 95% exact binomial confidence interval.
Progression free survival (PFS) | From start of protocol treatment to disease relapse/progression or death due to any cause, whichever is earlier, assessed up to 2 years
  PFS will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error; 95% confidence interval will be constructed based on log-log transformation. Median PFS will be estimated when possible.
Duration of response (DOR) | From the first achievement of CR or PR to disease progression/relapse or death due to any cause, whichever is earlier, assessed up to 2 years
  Response will be graded by the Lugano 2016 criteria. DOR will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error; 95% confidence interval will be constructed based on log-log transformation. Median DOR will be estimated when possible.

CONTACTS AND LOCATIONS:
Overall Officials: Swetha Kambhampati, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - City of Hope at Irvine Lennar, Irvine, California